CLINICAL TRIAL: NCT01976949
Title: Evaluation of a Social-networking Intervention to Reduce Cancer-related Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jason Owen, Phd., Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 57065; PA06-225 (Other Grant/Funding Number: Funding Opportunity Number)
Record Dates: First submitted 2013-09-24; First posted 2013-11-06 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Cancer Survivors With Clinically Significant Distress
Keywords: Cancer, social-networking intervention, cancer-related distress, internet health services, intervention delivery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Social-networking intervention (Active Comparator): Individuals interested in participating in the study will be randomized to receive access to a 12-week internet-based treatment group. Subjects assigned to the treatment group will have access to a group discussion board, a structured 12-week coping-skills training course, professional facilitation of the group, a real-time chat board, and personal profiles established by other group members. Subjects will be asked to complete online self-report measures of distress, mood disturbance, and quality of life at baseline and again after participation in the 12-week group.
  Interventions: Behavioral: online social-networking intervention
- Control group (Active Comparator): 12 week wait-list control subjects will be able to join a group after they complete the 12-week assessment and will be asked to complete a 24-week assessment in order to measure change over time. Subjects will have access to a group discussion board, a structured 12-week coping-skills training course, professional facilitation of the group, a real-time chat board, and personal profiles established by other group members. Subjects will be asked to complete online self-report measures of distress, mood disturbance, and quality of life at baseline and again after participation in the 12-week group.
  Interventions: Behavioral: online social-networking intervention

INTERVENTIONS:
Behavioral: online social-networking intervention

SUMMARY:
It is hypothesized that the treatment group will show greater improvements in quality of life and mood disturbance compared to the control group and that greater levels of engagement with the intervention materials will be associated with greater improvements in mood and quality of life.

DETAILED DESCRIPTION:
Individuals with cancer face an array of psychosocial needs, and it has been estimated that up to 35% of cancer survivors experience clinically-significant levels of distress. Psychosocial interventions may be effective for improving quality of life and reducing levels of mood disturbance in these patients. Unfortunately, barriers to accessing psychosocial intervention are common, and many are unable to access those services. Internet- based psychosocial interventions improve accessibility of care and offer additional methodological advantages, including the ability to easily collect self-report data, track exposure to the intervention, and evaluate effects of specific intervention components. The proposed study will evaluate whether a website developed specifically for providing psychological treatment and enhancing communication between cancer survivors can improve distress among cancer survivors who indicate that they have high levels of distress. If successful, the study will also provide valuable information needed to improve the treatment and to adequately conduct a larger trial comparing internet-based and face-to-face treatments.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age,
2. previous cancer diagnosis other than non-melanoma skin cancer,

4) fluent in English, 5) routine access to the Internet, and 6) presence of greater than mild distress as identified by having distress greater than or equal to 4 on initial screening with the Distress Thermometer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in -Overall Psychological Functioning (OQ-45) | 3-month change
  The OQ-45 measures the global functioning of a client and is composed of 3 subscales that measure subjective discomfort (intrapsychic functioning), interpersonal relationships, and social role performance. The OQ-45 has adequate internal consistency (a = .93) and reliability (r = .84) (Lambert, et al., 2004).
Change in-Center for Epidemiologic Studies Depress (CES-D) scale | 3-month change
  The CES-D is a self-report measure that consists of 20 items rated on a 4-point Likert scale to assess depressive symptoms experienced in the previous week. The CES-D has demonstrated excellent reliability and validity (Radloff, 1977). The standard cutoff score of 16 will be used to identify depression.
Anxiety | 3-month change
  Anxiety subscale of the brief Profile of Mood States (b-POMS; Shacham, 1983), which utilizes 37 descriptive mood adjectives to describe how a participant felt during the past week on a 5-point Likert scale. Specifically look at anxiety (anx subscale of POMS), vigor (subscale of POMS), and fatigue (subscale of POMS).

SECONDARY OUTCOMES:
Fatigue | 3-month change
  Fatigue subscale of the Profile of Mood States questionnaire
Vigor | 3-month change
  Vigor subscale of the Profile of Mood States questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jason E Owen, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

REFERENCES:
- [Background] Allen SM, Shah AC, Nezu AM, Nezu CM, Ciambrone D, Hogan J, Mor V. A problem-solving approach to stress reduction among younger women with breast carcinoma: a randomized controlled trial. Cancer. 2002 Jun 15;94(12):3089-100. doi: 10.1002/cncr.10586. PMID 12115339
- [Background] Austenfeld JL, Stanton AL. Coping through emotional approach: a new look at emotion, coping, and health-related outcomes. J Pers. 2004 Dec;72(6):1335-63. doi: 10.1111/j.1467-6494.2004.00299.x. PMID 15509285
- [Background] Baker F, Denniston M, Zabora J, Polland A, Dudley WN. A POMS short form for cancer patients: psychometric and structural evaluation. Psychooncology. 2002 Jul-Aug;11(4):273-81. doi: 10.1002/pon.564. PMID 12203741
- [Background] Bantum EO, Owen JE. Evaluating the validity of computerized content analysis programs for identification of emotional expression in cancer narratives. Psychol Assess. 2009 Mar;21(1):79-88. doi: 10.1037/a0014643. PMID 19290768
- [Background] Beskow LM, Sandler RS, Weinberger M. Research recruitment through US central cancer registries: balancing privacy and scientific issues. Am J Public Health. 2006 Nov;96(11):1920-6. doi: 10.2105/AJPH.2004.061556. Epub 2006 Mar 29. PMID 16571700
- [Background] Beskow LM, Millikan RC, Sandler RS, Godley PA, Weiner BJ, Weinberger M. The effect of physician permission versus notification on research recruitment through cancer registries (United States). Cancer Causes Control. 2006 Apr;17(3):315-23. doi: 10.1007/s10552-005-0521-1. PMID 16489539
- [Background] Brooks R. EuroQol: the current state of play. Health Policy. 1996 Jul;37(1):53-72. doi: 10.1016/0168-8510(96)00822-6. PMID 10158943
- [Background] Carlson LE, Angen M, Cullum J, Goodey E, Koopmans J, Lamont L, MacRae JH, Martin M, Pelletier G, Robinson J, Simpson JS, Speca M, Tillotson L, Bultz BD. High levels of untreated distress and fatigue in cancer patients. Br J Cancer. 2004 Jun 14;90(12):2297-304. doi: 10.1038/sj.bjc.6601887. PMID 15162149
- [Background] Carmack Taylor CL, Kulik J, Badr H, Smith M, Basen-Engquist K, Penedo F, Gritz ER. A social comparison theory analysis of group composition and efficacy of cancer support group programs. Soc Sci Med. 2007 Jul;65(2):262-73. doi: 10.1016/j.socscimed.2007.03.024. Epub 2007 Apr 19. PMID 17448580
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Cheshire C, Antin A. (2008). The social psychological effects of feedback on the production of Internet information pools. J Computer-Mediated Communication, 13, 705-27.
- [Background] Cunningham AJ, Edmonds CV, Jenkins GP, Pollack H, Lockwood GA, Warr D. A randomized controlled trial of the effects of group psychological therapy on survival in women with metastatic breast cancer. Psychooncology. 1998 Nov-Dec;7(6):508-17. doi: 10.1002/(SICI)1099-1611(199811/12)7:63.0.CO;2-7. PMID 9885092
- [Background] Edwards AG, Hailey S, Maxwell M. Psychological interventions for women with metastatic breast cancer. Cochrane Database Syst Rev. 2004;(2):CD004253. doi: 10.1002/14651858.CD004253.pub2. PMID 15106244
- [Background] Erdfelder E, Faul F, Buchner A. (1996). G*Power: A general power analysis program. Behavior Research, Methods, Instruments, and Computers, 28, 1-11.
- [Background] Fawzy FI, Fawzy NW. A structured psychoeducational intervention for cancer patients. Gen Hosp Psychiatry. 1994 May;16(3):149-92. doi: 10.1016/0163-8343(94)90098-1. No abstract available. PMID 8063085
- [Background] Folkman S, Greer S. Promoting psychological well-being in the face of serious illness: when theory, research and practice inform each other. Psychooncology. 2000 Jan-Feb;9(1):11-9. doi: 10.1002/(sici)1099-1611(200001/02)9:13.0.co;2-z. PMID 10668055
- [Background] Fonteyn M, Bauer-Wu S. Using qualitative evaluation in a feasibility study to improve and refine a complementary therapy intervention prior to subsequent research. Complement Ther Clin Pract. 2005 Nov;11(4):247-52. doi: 10.1016/j.ctcp.2005.05.007. Epub 2005 Nov 2. PMID 16290895
- [Background] Fukui S, Kugaya A, Kamiya M, Koike M, Okamura H, Nakanishi T, Wenner M, Imoto S, Kanagawa K, Uchitomi Y. Participation in psychosocial group intervention among Japanese women with primary breast cancer and its associated factors. Psychooncology. 2001 Sep-Oct;10(5):419-27. doi: 10.1002/pon.534. PMID 11536420
- [Background] Ganz PA, Kwan L, Stanton AL, Krupnick JL, Rowland JH, Meyerowitz BE, Bower JE, Belin TR. Quality of life at the end of primary treatment of breast cancer: first results from the moving beyond cancer randomized trial. J Natl Cancer Inst. 2004 Mar 3;96(5):376-87. doi: 10.1093/jnci/djh060. PMID 14996859
- [Background] Graves KD. Social cognitive theory and cancer patients' quality of life: a meta-analysis of psychosocial intervention components. Health Psychol. 2003 Mar;22(2):210-9. PMID 12683741
- [Background] Gustafson DH, Wise M, McTavish F, et al. (1993). Development and pilot evaluation of a computer-based support system for women with breast cancer. J Psychosoc Oncol, 11, 69-93.
- [Background] Gustafson DH, McTavish F, Hawkins R, Pingree S, Arora N, Mendenhall J, Simmons GE. Computer support for elderly women with breast cancer. JAMA. 1998 Oct 21;280(15):1305. doi: 10.1001/jama.280.15.1305. No abstract available. PMID 9794300
- [Background] Gustafson DH, Hawkins R, Pingree S, McTavish F, Arora NK, Mendenhall J, Cella DF, Serlin RC, Apantaku FM, Stewart J, Salner A. Effect of computer support on younger women with breast cancer. J Gen Intern Med. 2001 Jul;16(7):435-45. doi: 10.1046/j.1525-1497.2001.016007435.x. PMID 11520380
- [Background] Gustafson DH, Hawkins RP, Boberg EW, McTavish F, Owens B, Wise M, Berhe H, Pingree S. CHESS: 10 years of research and development in consumer health informatics for broad populations, including the underserved. Int J Med Inform. 2002 Nov 12;65(3):169-77. doi: 10.1016/s1386-5056(02)00048-5. PMID 12414016
- [Background] Hann D, Winter K, Jacobsen P. Measurement of depressive symptoms in cancer patients: evaluation of the Center for Epidemiological Studies Depression Scale (CES-D). J Psychosom Res. 1999 May;46(5):437-43. doi: 10.1016/s0022-3999(99)00004-5. PMID 10404478
- [Background] Hartoonian N, Ormseth S, Bantum EO, Owen JE. (2008). Process and outcome evaluation of a social- networking website for health promotion. Ann Behav Med, 35s, 63.
- [Background] Helgeson VS, Cohen S, Schulz R, Yasko J. Group support interventions for women with breast cancer: who benefits from what? Health Psychol. 2000 Mar;19(2):107-14. doi: 10.1037//0278-6133.19.2.107. PMID 10762094
- [Background] Helgeson VS, Lepore SJ, Eton DT. Moderators of the benefits of psychoeducational interventions for men with prostate cancer. Health Psychol. 2006 May;25(3):348-54. doi: 10.1037/0278-6133.25.3.348. PMID 16719606
- [Background] Hewitt M, Rowland JH. Mental health service use among adult cancer survivors: analyses of the National Health Interview Survey. J Clin Oncol. 2002 Dec 1;20(23):4581-90. doi: 10.1200/JCO.2002.03.077. PMID 12454116
- [Background] Hilarius DL, Kloeg PH, Detmar SB, Muller MJ, Aaronson NK. Level of agreement between patient self-report and observer ratings of health-related quality of life communication in oncology. Patient Educ Couns. 2007 Jan;65(1):95-100. doi: 10.1016/j.pec.2006.06.002. Epub 2006 Jul 26. PMID 16872790
- [Background] Hsu J, Huang J, Kinsman J, Fireman B, Miller R, Selby J, Ortiz E. Use of e-Health services between 1999 and 2002: a growing digital divide. J Am Med Inform Assoc. 2005 Mar-Apr;12(2):164-71. doi: 10.1197/jamia.M1672. Epub 2004 Nov 23. PMID 15561786
- [Background] Institute of Medicine (US) and National Research Council (US) National Cancer Policy Board; Hewitt M, Herdman R, Holland J, editors. Meeting Psychosocial Needs of Women with Breast Cancer. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK215943/ PMID 25009861
- [Background] Jacobsen PB, Meade CD, Stein KD, Chirikos TN, Small BJ, Ruckdeschel JC. Efficacy and costs of two forms of stress management training for cancer patients undergoing chemotherapy. J Clin Oncol. 2002 Jun 15;20(12):2851-62. doi: 10.1200/JCO.2002.08.301. PMID 12065562
- [Background] Jacobsen PB, Donovan KA, Trask PC, Fleishman SB, Zabora J, Baker F, Holland JC. Screening for psychologic distress in ambulatory cancer patients. Cancer. 2005 Apr 1;103(7):1494-502. doi: 10.1002/cncr.20940. PMID 15726544
- [Background] Jacobsen P, Donovan K, Swaine Z, Watson I. (2006). Management of anxiety and depression in adult cancer patients: Toward an evidence-based approach. In Oncology: An evidence-based approach. A. Chang, P. Ganz, D. Hayes, T. Kinsella, H. Pass, J. Schiller, R. Stone, V. Strecher (Eds.). New York: Springer-Verlag, p. 1552-1579.
- [Background] Kwekkeboom KL. Outcome expectancy and success with cognitive-behavioral interventions: the case of guided imagery. Oncol Nurs Forum. 2001 Aug;28(7):1125-32. PMID 11517846
- [Background] Lazarus RS, Folkman S. (1984). Stress, appraisal, and coping. New York: Springer.
- [Background] Lee V, Robin Cohen S, Edgar L, Laizner AM, Gagnon AJ. Meaning-making intervention during breast or colorectal cancer treatment improves self-esteem, optimism, and self-efficacy. Soc Sci Med. 2006 Jun;62(12):3133-45. doi: 10.1016/j.socscimed.2005.11.041. Epub 2006 Jan 18. PMID 16413644
- [Background] Lieberman MA, Golant M, Giese-Davis J, Winzlenberg A, Benjamin H, Humphreys K, Kronenwetter C, Russo S, Spiegel D. Electronic support groups for breast carcinoma: a clinical trial of effectiveness. Cancer. 2003 Feb 15;97(4):920-5. doi: 10.1002/cncr.11145. PMID 12569591
- [Background] Liess A, Simon W, Yutsis M, Owen JE, Piemme KA, Golant M, Giese-Davis J. Detecting emotional expression in face-to-face and online breast cancer support groups. J Consult Clin Psychol. 2008 Jun;76(3):517-23. doi: 10.1037/0022-006X.76.3.517. PMID 18540745
- [Background] Badia Llach X, Herdman M, Schiaffino A. Determining correspondence between scores on the EQ-5D "thermometer" and a 5-point categorical rating scale. Med Care. 1999 Jul;37(7):671-7. doi: 10.1097/00005650-199907000-00007. PMID 10424638
- [Background] Meyer TJ, Mark MM. Effects of psychosocial interventions with adult cancer patients: a meta-analysis of randomized experiments. Health Psychol. 1995 Mar;14(2):101-8. doi: 10.1037//0278-6133.14.2.101. PMID 7789344
- [Background] Newell SA, Sanson-Fisher RW, Savolainen NJ. Systematic review of psychological therapies for cancer patients: overview and recommendations for future research. J Natl Cancer Inst. 2002 Apr 17;94(8):558-84. doi: 10.1093/jnci/94.8.558. PMID 11959890
- [Background] Nezu AM, Nezu CM, Friedman SH, Faddis S, Houts PS. (1998). Helping cancer patients cope: A problem- solving approach. Washinton, D.C.: American Psychological Association.
- [Background] Overcash J, Extermann M, Parr J, Perry J, Balducci L. Validity and reliability of the FACT-G scale for use in the older person with cancer. Am J Clin Oncol. 2001 Dec;24(6):591-6. doi: 10.1097/00000421-200112000-00013. PMID 11801761
- [Background] Owen JE, Klapow JC, Hicken B, Tucker DC. Psychosocial interventions for cancer: review and analysis using a three-tiered outcomes model. Psychooncology. 2001 May-Jun;10(3):218-30. doi: 10.1002/pon.509. PMID 11351374
- [Background] Owen JE, Yarbrough EJ, Vaga A, Tucker DC. (2003). Investigation of the effects of gender and preparation on quality of communication in Internet support groups. Comp Hum Behav, 19, 259-75.
- [Background] Owen JE, Klapow JC, Roth DL, Nabell L, Tucker DC. Improving the effectiveness of adjuvant psychological treatment for women with breast cancer: the feasibility of providing online support. Psychooncology. 2004 Apr;13(4):281-92. doi: 10.1002/pon.733. PMID 15054732
- [Background] Owen JE, Klapow JC, Roth DL, Shuster JL Jr, Bellis J, Meredith R, Tucker DC. Randomized pilot of a self-guided internet coping group for women with early-stage breast cancer. Ann Behav Med. 2005 Aug;30(1):54-64. doi: 10.1207/s15324796abm3001_7. PMID 16097906
- [Background] Owen JE, Giese-Davis J, Cordova M, Kronenwetter C, Golant M, Spiegel D. Self-report and linguistic indicators of emotional expression in narratives as predictors of adjustment to cancer. J Behav Med. 2006 Aug;29(4):335-45. doi: 10.1007/s10865-006-9061-8. Epub 2006 Jul 15. PMID 16845583
- [Background] Owen JE, Goldstein MS, Lee JH, Breen N, Rowland JH. Use of health-related and cancer-specific support groups among adult cancer survivors. Cancer. 2007 Jun 15;109(12):2580-9. doi: 10.1002/cncr.22719. PMID 17503435
- [Background] Pennebaker JW, Francis ME. (2001). Linguistic Inquiry and Word Count. Mahwah, NJ Erlbaum.
- [Background] Pew Internet and American Life Project (2003). How Californians compare to the rest of the nation. PIP: Washington, D.C.
- [Background] Pew Internet & American Life Project. (2007). E-patients with a disability or chronic disease. http://www.pewinternet.org/pdfs/EPatients_Chronic_Conditions_2007.pdf, last accessed on 1/16/08.
- [Background] Radloff LS. (1977). The CES-D scale: A self-report depression scale for research in the general population. App Psychol Measures, 1, 385-401.
- [Background] Rehse B, Pukrop R. Effects of psychosocial interventions on quality of life in adult cancer patients: meta analysis of 37 published controlled outcome studies. Patient Educ Couns. 2003 Jun;50(2):179-86. doi: 10.1016/s0738-3991(02)00149-0. PMID 12781933
- [Background] Roth AJ, Kornblith AB, Batel-Copel L, Peabody E, Scher HI, Holland JC. Rapid screening for psychologic distress in men with prostate carcinoma: a pilot study. Cancer. 1998 May 15;82(10):1904-8. doi: 10.1002/(sici)1097-0142(19980515)82:103.0.co;2-x. PMID 9587123
- [Background] Shacham S. A shortened version of the Profile of Mood States. J Pers Assess. 1983 Jun;47(3):305-6. doi: 10.1207/s15327752jpa4703_14. PMID 6886962
- [Background] Spiegel D, Classen C. (2000). Group therapy for cancer patients: A research-based handbook of psychosocial care. New York: Basic Books.
- [Background] Stanton AL, Kirk SB, Cameron CL, Danoff-Burg S. Coping through emotional approach: scale construction and validation. J Pers Soc Psychol. 2000 Jun;78(6):1150-69. doi: 10.1037//0022-3514.78.6.1150. PMID 10870915
- [Background] Stanton AL, Danoff-Burg S, Sworowski LA, Collins CA, Branstetter AD, Rodriguez-Hanley A, Kirk SB, Austenfeld JL. Randomized, controlled trial of written emotional expression and benefit finding in breast cancer patients. J Clin Oncol. 2002 Oct 15;20(20):4160-8. doi: 10.1200/JCO.2002.08.521. PMID 12377959
- [Background] Vilela LD, Nicolau B, Mahmud S, Edgar L, Hier M, Black M, Franco EL, Allison PJ. Comparison of psychosocial outcomes in head and neck cancer patients receiving a coping strategies intervention and control subjects receiving no intervention. J Otolaryngol. 2006 Apr;35(2):88-96. doi: 10.2310/7070.2005.5002. PMID 16527026
- [Background] Watts S, Edgar L. Nucare, a coping skills training intervention for oncology patients and families: participants' motivations and expectations. Can Oncol Nurs J. 2004 Spring;14(2):84-95. English, French. PMID 15230029
- [Background] Weiss D, Marmar C. (1997). The Impact of Event Scale - Revised. In J. Wilson & T. Keane (Eds), Assessing psychological trauma and PTSD. New York: Guilford Press.
- [Background] Winzelberg AJ, Classen C, Alpers GW, Roberts H, Koopman C, Adams RE, Ernst H, Dev P, Taylor CB. Evaluation of an internet support group for women with primary breast cancer. Cancer. 2003 Mar 1;97(5):1164-73. doi: 10.1002/cncr.11174. PMID 12599221
- [Background] Zabora J, BrintzenhofeSzoc K, Curbow B, Hooker C, Piantadosi S. The prevalence of psychological distress by cancer site. Psychooncology. 2001 Jan-Feb;10(1):19-28. doi: 10.1002/1099-1611(200101/02)10:13.0.co;2-6. PMID 11180574
- [Derived] Owen JE, O'Carroll Bantum E, Pagano IS, Stanton A. Randomized Trial of a Social Networking Intervention for Cancer-Related Distress. Ann Behav Med. 2017 Oct;51(5):661-672. doi: 10.1007/s12160-017-9890-4. PMID 28244002
- See also: Study website — http://www.health-space.net